CLINICAL TRIAL: NCT04462978
Title: Investigating Clinical Features, Natural Course and Pathophysiology of Non-Immunoglobulin E-mediated Food Allergies in the Pediatric Age
Brief Title: Non-Immunoglobulin E-mediated Food Allergies in Children
Acronym: NIGEFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Professor of Pediatrics, Federico II University
Other Study IDs: 102/20
Record Dates: First submitted 2020-05-28; First posted 2020-07-08 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Non IgE Mediated Food Allergy; Food Protein-Induced Enteropathy; Food Protein-Induced Proctocolitis; Food Protein-Induced Enterocolitis Syndrome; Food Protein-induced Motility Disorders
Keywords: Food allergy; Adverse food reactions; Immune tolerance; Atopy patch test; Atopic march; Oral food challenge; Food Protein-Induced Enteropathy; Food Protein-Induced Proctocolitis; Food Protein-Induced Enterocolitis Syndrome; Food protein-induced motility disorders
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples Peripheral blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non IgE-mediated food allergy: Children with non IgE-mediated food allergy
  Interventions: Other: Non IgE-mediated food allergy

INTERVENTIONS:
Other: Non IgE-mediated food allergy

SUMMARY:
Non-IgE-mediated gastrointestinal food allergies (non-IgE-GIFA) are an evolving web of clinical conditions characterized by subacute and/or chronic symptoms and include food protein-induced enterocolitis syndrome (FPIES), food protein-induced enteropathy (FPE), food protein-induced allergic proctocolitis (FPIAP), and food protein-induced allergic dysmotility disorders (gastroesophageal reflux disease (GERD), colic and constipation) (FPIMD).

Despite the prevalence and clinical impact of these conditions, the pathogenesis as well as the natural history and the best management of these disorders are still poorly defined. These limitations could be responsible for diagnostic delays and errors, and suboptimal clinical management. We aim to evaluate clinical features, natural course and pathophysiology of non-IgE-GIFA in the pediatric age.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged between 0-14 years
* suggestive history of food allergy

Exclusion Criteria:

* age >14 years-
* chronic systemic diseases,
* malignancy,
* immunodeficiency,
* infectious diseases,
* autoimmune diseases,
* inflammatory bowel diseases,
* celiac disease,
* metabolic and genetic diseases,
* cystic fibrosis,
* chronic pulmonary diseases,
* gastrointestinal, respiratory, urinary tract and/or cardiovascular malformations,
* neurologic and/or neuropsychiatric disorders,
* gastrointestinal tract eosinophilic disorders,
* use of immunomodulating drugs, steroids, pre-pro-synbiotics, antibiotics in the previous 4 months

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: subjects consecutively observed at the Pediatric Allergy Program, at the Department of Translational Medical Science of the University of Naples Federico II, both sex, aged between 0-14 years with suggestive history of food allergy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical features and disease course of non-IgE mediated food allergies in children | After 72 months from the study start
  Rate of pts affected by FPIES, FPE, FPIAP, FPIMD; diagnostic delay; disease duration, rate of pts with mono vs poli food allergies; main antigens responsible for the diseases; occurrence of atopic dermatitis before food allergy onset; results of allergy screening tests; occurrence of atopic march
Evaluation of clinical features of non-IgE mediated food allergies in children | After 72 months from the study start
  Dietary management and Nutritional status (weight and height will be combined to report BMI z-score)

SECONDARY OUTCOMES:
Evaluation of immune mechanisms involved in the pathogenesis of non-IgE mediated food allergies in children | through study completion, an average of 2 years
  Evaluation of serum levels of Th2, Th1, and Th17 cytokines
Evaluation of immune mechanisms involved in the pathogenesis of non-IgE mediated food allergies in children | through study completion, an average of 2 years
  Evaluation of epigenetic mechanisms
Evaluation of immune mechanisms involved in the pathogenesis of non-IgE mediated food allergies in children | through study completion, an average of 2 years
  Evaluation of immune cells phenotype
Evaluation of immune mechanisms involved in the pathogenesis of non-IgE mediated food allergies in children | through study completion, an average of 2 years
  Evaluation of mithocondrial metabolism of human lymphocytes
Evaluation of gut microbiome features in children with Non-IgE-mediated food allergies | through study completion, an average of 2 years
  Evaluation of gut microbiome structure and function

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided